CLINICAL TRIAL: NCT07391137
Title: The Effects of a Dietary Regimen Characterized by High Consumption of Cruciferous Vegetables on Recurrence-free Survival in Patients With Intermediate, High and Very High-risk Non-Muscle Invasive Bladder Cancer: a Randomized Trial
Brief Title: CRUCIAL-R Study : Cruciferous Vegetables Dietary Regimen in NMIBC
Acronym: CRUCIAL-R
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: S. Andrea Hospital (Other)
Responsible Party: Principal Investigator, Cosimo De Nunzio, P.I. Professor, S. Andrea Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CRUCIAL-R
Record Dates: First submitted 2025-04-15; First posted 2026-02-05 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Recurrence Free Survival; Bladder Cancer Recurrence
Keywords: Bladder Cancer; NMIBC; Cruciferae; recurrence
MeSH Terms: conditions — Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Neoplasms; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 - Patients with Cruciferae intake diet (Experimental): Patients with Cruciferae intake diet
  Interventions: Dietary Supplement: Cruciferae intake diet
- 2 (Placebo Comparator): Patients with normal diet
  Interventions: Dietary Supplement: Habituary dietary regimen

INTERVENTIONS:
Dietary Supplement: Cruciferae intake diet — Patients in the intervention group will receive a dietary regimen characterized by high consumption of Cruciferae vegetables [≥1 cup /day] for 6 months. Patients in this group will receive educative booklets on the Cruciferae family of vegetables and visual charts on serving sizing to meet the recommended daily CV intake. Patients will be asked to record daily Cruciferae intake. They will receive a live phone call every week to verify their understanding of the educational information and the consistency of the dietary regimen.
  Arms: 1 - Patients with Cruciferae intake diet
Dietary Supplement: Habituary dietary regimen — Patients randomized in the control group will receive standard of care (SOC) without any modification of the habitual dietary regimen.
  Arms: 2

SUMMARY:
Emerging evidence highlights the importance of nutrition in modulating cancer-related pathways, suggesting that specific dietary patterns and food choices may influence cancer risk. A protective role has been suggested for high consumption of vegetables, non-saturated fat oil (Mediterranean diet), fruits, and flavonoids [10-13]. In contrast, a diet rich in saturated fats and meat has been linked to an increased risk of BC [14,15]. Particularly, the consumption of vegetables of the Cruciferae family, such as broccoli, cauliflower, brussels sprouts, cabbage, kale, turnips, and others, has gathered attention for their potential protective effects due to their bioactive compounds: Isothiocyanates (ITCs). Dietary ITCs are a group of phytochemicals with multifaceted anticancer mechanisms primarily derived from cruciferous vegetables (CV) as glucosinolates and converted to ITCs by the action of the enzyme myrosinase [16]. Organic ITCs, particularly allyl isothiocyanate (AITC), benzyl isothiocyanate (BITC), phenethyl isothiocyanate (PEITC), and sulforaphane (SF), are among the most extensively studied cancer chemopreventive agents. Several mechanisms for ITCs in protection against carcinogenesis have been proposed, which include inhibition of carcinogen activation and promotion of detoxification, induction of cell cycle arrest and activation of apoptosis, inhibition of cancer cell invasion, modulation of the tumor microenvironment, inhibition of self-renewal of stem cells, rearrangement of energy metabolism and regulation of microbial homeostasis [17-22].

Aims Primary Objective

• To evaluate the effect, in terms of recurrence-free survival (RFS) at 1 year, of a dietary regimen characterized by high consumption of the Cruciferae family vegetables versus no dietary regimen in patients with Intermediate, High, or Very High-grade Non-Muscle Invasive Bladder Cancer treated with BCG (defined as the standard of care - SOC).

Secondary Objectives

* To evaluate the effect, in terms of time to recurrence, of a dietary regimen characterized by high consumption of the Cruciferae family vegetables versus no dietary regimen in patients with Intermediate, High, and Very High-grade Non-Muscle Invasive Bladder Cancer.
* To evaluate the effect, in terms of recurrence-free survival (RFS), of a dietary regimen characterized by high consumption of the Cruciferae family vegetables versus no dietary regimen in patients with Intermediate, High, and Very High-grade Non-Muscle Invasive Bladder Cancer with prior recurrence ≤1/yr and <4 tumors (according to 2016 EORTC risk stratification for patients treated with maintenance BCG).
* To evaluate the impact of high Cruciferous vegetable consumption on urinary ITC levels.
* To evaluate the impact of high Cruciferous vegetable consumption on quality of life (QoL).

DETAILED DESCRIPTION:
Background Bladder cancer (BC) ranks as the seventh most common cancer among men globally and the tenth when both genders are considered. The majority (up to 75%) of newly diagnosed BC presents as non-muscle-invasive BC (NMIBC) including Ta (non-invasive papillary carcinoma confined to the mucosa), CIS (Carcinoma in Situ, a flat, high grade, non-invasive urothelial carcinoma) and T1 (tumor invasion of the sub-epithelial connective tissue) disease stage. NMIBC has a high prevalence due to low progression rates and long-term survival, representing a significant burden on both public health and individual well-being. The prevalence of urothelial BC is among the highest for all urologic malignancies. Although the understanding of genetic susceptibility is growing steadily, no clinically relevant genetic alteration has been linked to BC up to date, and family history seems to have little impact on BC risk. Conversely, most BC cases are associated with external exposure to carcinogens. Supportive evidence has been reported on several risk factors: tobacco smoking alone accounts for approximately 50% of events. In contrast, occupational exposure (mostly involving aromatic amines, polycyclic, and chlorinated hydrocarbons) represents the second most common risk factor in industrialized countries. Environmental exposure (e.g., trihalomethanes and arsenic in drinking water) and pelvic radiation have been linked to an increased risk of developing BC. In light of the significant impact of modifiable risk factors on the incidence of BC, implementation of primary prevention strategies can lead to a decrease in BC risk: in the "Women's Health Initiative (WHI) Study" a decrease in BC risk was demonstrated after smoking cessation. Likewise, work-safety guidelines have been prompted to reduce the extent of professional exposure in developed industrial settings, thus eliminating the difference in BC incidence between chemical workers and the general population. Primary interventions targeting exposure and lifestyle changes have become central to public health strategies aimed at mitigating the burden of bladder cancer. In the broader landscape of primary prevention, dietary habits play a crucial role in reducing the risk of bladder cancer. Emerging evidence highlights the importance of nutrition in modulating cancer-related pathways, suggesting that specific dietary patterns and food choices may influence cancer risk. A protective role has been suggested for high consumption of vegetables, non-saturated fat oil (Mediterranean diet), fruits, and flavonoids. In contrast, a diet rich in saturated fats and meat has been linked to an increased risk of BC. Particularly, the consumption of vegetables of the Cruciferae family, such as broccoli, cauliflower, brussels sprouts, cabbage, kale, turnips, and others, has gathered attention for their potential protective effects due to their bioactive compounds: Isothiocyanates (ITCs). Dietary ITCs are a group of phytochemicals with multifaceted anticancer mechanisms primarily derived from cruciferous vegetables (CV) as glucosinolates and converted to ITCs by the action of the enzyme myrosinase. Organic ITCs, particularly allyl isothiocyanate (AITC), benzyl isothiocyanate (BITC), phenethyl isothiocyanate (PEITC), and sulforaphane (SF), are among the most extensively studied cancer chemopreventive agents. Several mechanisms for ITCs in protection against carcinogenesis have been proposed, which include inhibition of carcinogen activation and promotion of detoxification, induction of cell cycle arrest and activation of apoptosis, inhibition of cancer cell invasion, modulation of the tumor microenvironment, inhibition of self-renewal of stem cells, rearrangement of energy metabolism and regulation of microbial homeostasis. Several in vitro, in vivo, and epidemiologic studies have shown that a diet rich in vegetables in the Cruciferae family may lower overall cancer risk for breast, colorectal, lung, and prostate cancer. The important role of dietary ITCs has been demonstrated in reducing BC risk and BC-specific mortality. In vitro, the 4 most common dietary ITCs and their primary urinary metabolites showed inhibition of growth of a panel of human bladder cancer cells, including NMIBC cells, with half-maximal inhibitory concentration (IC50) values around 10 µmol on average, which is achievable in the urine with a single oral dose of ITC at 10 µmol/kg in rats, also readily achievable in humans, considering an average total isothiocyanate yield in Cruciferae of 16.2 μmol/100g wet weight. By increasing Cruciferae intake by 1 cup a day, the urinary concentration of ITCs increases on average by 10.4 µmol, the desirable dose level of urinary ITCs needed to stop or kill at least 50% of bladder cancer cells in in vitro models. Orally ingested ITCs are rapidly and almost exclusively delivered to the bladder and concentrated in the urine, showing concentration 2 or 3 times higher in the urine than in the plasma within 3 hours of dosing. This unique in vivo metabolism and disposition pathway renders the bladder the best target for ITCs' anticancer potential. In the Bladder Cancer Epidemiology, Wellness, and Lifestyle Study (Be-Well study), a multicenter prospective cohort study on newly diagnosed NMIBC, a possible beneficial role of dietary ITCs in NMIBC prognosis was assessed: despite no overall association between dietary ITC intake and recurrence risk was found, high ITC intake was linked to over twice the odds of late recurrence, while high raw cruciferous vegetable intake reduced the odds of multiple recurrences by 50%-60%, and elevated BITC and PEITC biomarkers were associated with >50% lower risk of muscle-invasive progression. In the same study group, the impact of dietary ITC exposure was assessed in relation to the efficacy of intravesical Mitomycin (MMC) chemotherapy or Bacillus Calmette-Guérin (BCG) immunotherapy on the risk of recurrence. In a stratified analysis, patients who received BCG and consumed high amounts (>2.4 servings/month with 1 serving corresponding to half a cup of non-leafy vegetables or 1 cup of leafy vegetables) of raw CVs had at least a 44% reduced risk of recurrence and multiple recurrences, which was not observed in those consuming low doses of row CV. In a randomized controlled setting, this study aims to assess the impact of CV intake and ITC exposure on recurrence risk in patients with NMIBC undergoing BCG intravesical immunotherapy.

Hypothesis Primary interventions targeting exposure and lifestyle changes have become central to public health strategies aimed at mitigating the burden of bladder cancer. In the broader landscape of primary prevention, dietary habits play a crucial role in reducing the risk of bladder cancer. Emerging evidence highlights the importance of nutrition in modulating cancer-related pathways, suggesting that specific dietary patterns and food choices may influence cancer risk. A protective role has been suggested for high consumption of vegetables, non-saturated fat oil (Mediterranean diet), fruits, and flavonoids. In contrast, a diet rich in saturated fats and meat has been linked to an increased risk of BC. Particularly, the consumption of vegetables of the Cruciferae family, such as broccoli, cauliflower, brussels sprouts, cabbage, kale, turnips, and others, has gathered attention for their potential protective effects due to their bioactive compounds: Isothiocyanates (ITCs). Dietary ITCs are a group of phytochemicals with multifaceted anticancer mechanisms primarily derived from cruciferous vegetables (CV) as glucosinolates and converted to ITCs by the action of the enzyme myrosinase. Organic ITCs, particularly allyl isothiocyanate (AITC), benzyl isothiocyanate (BITC), phenethyl isothiocyanate (PEITC), and sulforaphane (SF), are among the most extensively studied cancer chemopreventive agents. Several mechanisms for ITCs in protection against carcinogenesis have been proposed, which include inhibition of carcinogen activation and promotion of detoxification, induction of cell cycle arrest and activation of apoptosis, inhibition of cancer cell invasion, modulation of the tumor microenvironment, inhibition of self-renewal of stem cells, rearrangement of energy metabolism and regulation of microbial homeostasis.

Aims Primary Objective

• To evaluate the effect, in terms of recurrence-free survival (RFS) at 1 year, of a dietary regimen characterized by high consumption of the Cruciferae family vegetables versus no dietary regimen in patients with Intermediate, High, or Very High-grade Non-Muscle Invasive Bladder Cancer treated with BCG (defined as the standard of care - SOC).

Secondary Objectives

* To evaluate the effect, in terms of time to recurrence, of a dietary regimen characterized by high consumption of the Cruciferae family vegetables versus no dietary regimen in patients with Intermediate, High, and Very High-grade Non-Muscle Invasive Bladder Cancer.
* To evaluate the effect, in terms of recurrence-free survival (RFS), of a dietary regimen characterized by high consumption of the Cruciferae family vegetables versus no dietary regimen in patients with Intermediate, High, and Very High-grade Non-Muscle Invasive Bladder Cancer with prior recurrence ≤1/yr and <4 tumors (according to 2016 EORTC risk stratification for patients treated with maintenance BCG).
* To evaluate the impact of high Cruciferous vegetable consumption on urinary ITC levels.
* To evaluate the impact of high Cruciferous vegetable consumption on quality of life (QoL).

Experimental design This study is a parallel-group, randomized controlled trial with a 1:1 allocation ratio designed to assess the superiority of a high-cruciferous vegetable dietary regimen compared to standard care in reducing bladder cancer recurrence.

Intervention The subjects will be assessed for eligibility at the screening visit (Visit 1) three weeks after TURB before randomization, and only subjects who fulfill the inclusion criteria will be included: patients with a diagnosis of Intermediate, High, and Very High-risk NMIBC, according to the new EAU NMIBC prognostic factor risk groups. Patients in the intervention group will receive a dietary regimen characterized by high consumption of Cruciferae vegetables [≥1 cup /day] for 6 months. Patients in this group will receive educative booklets on the Cruciferae family of vegetables and visual charts on serving sizing to meet the recommended daily CV intake. Patients will be asked to record daily Cruciferae intake. They will receive a live phone call every week to verify their understanding of the educational information and the consistency of the dietary regimen. Patients randomized in the control group will receive standard of care (SOC) without modifying the habitual nutritional regimen.

Study Timeline

Study Timeline Timepoint (mo) T0 1 2 3 4 5 6 7 8 9 10 11 12 ENROLMENT Eligibility screen X Informed Consent X Baseline clinical evaluation X Allocation X INTERVENTION Dietary Regimen vs SOC X X X X X X X ASSESSMENTS FU clinical evaluation X X X X FU phone call X X X X X X CLOSE-OUT X

Table 1. Study Timeline. Each participant will take part in the study for a total of 12 months after enrollment. Abbreviations: mo= months; FU= Follow-up.

Sample size A power analysis was conducted before data collection using SPSS to determine the appropriate sample size. A two-sided test with a Type I error rate (α) of 0.05 and a statistical power of 80% was performed to ensure adequate power for detecting a meaningful effect. The anticipated impact is the relative reduction of 40% (an absolute reduction of 10%) of the recurrence rate in the Study group versus the control group, given a recurrence rate in the general population (according to EAU risk stratification) of 25% at 1 year. To detect this difference, 250 patients per group are necessary, using the adjusted chi-square method.

Sequence generation and blinding The allocation sequence will be generated using computer-generated random numbers with a ratio of 1:1. This study will be conducted as an open-label trial. Due to the nature of the dietary intervention, neither participants nor study staff will be blinded to group assignment. However, outcome assessors analyzing urinary ITC levels and recurrence outcomes will be blinded to participant allocation.

Expected results The primary outcome of recurrence-free survival and the secondary outcome time to recurrence will be analyzed using Kaplan-Meier survival curves, and the intervention and control groups will be compared using the log-rank test. The Cox proportional hazards model will be applied to estimate hazard ratios, adjusting for relevant covariates such as age, gender, and baseline tumor characteristics. A two-tailed p-value < 0.05 will be considered statistically significant. Secondary outcomes, including urinary ITC levels, will be analyzed using t-tests or Mann-Whitney U tests for continuous variables and Chi-squared tests for categorical variables, depending on the data distribution. Descriptive statistics (mean, median, standard deviation) will be provided for all continuous variables and frequencies for categorical variables. A subgroup analysis will be conducted in subjects with prior recurrence ≤1/yr and <4 tumors (according to 2016 EORTC risk stratification for patients treated with maintenance BCG). An interim analysis will be conducted after 1 year of study enrollment to evaluate safety, efficacy, and trial progress.

Impact on cancer Low recurrence in bladder cancer

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed Non-Muscle Invasive Bladder Cancer of Intermediate, High, or Very High risk according to the 2021 EAU NMIBC scoring model.
* Age ≥ 18

Exclusion Criteria:

* Low-Risk Non-Muscle Invasive Bladder Cancer
* Muscle Invasive Bladder Cancer
* Life expectancy < 5 years
* WHO performance status 3 or 4
* Variant histology
* Concomitant Urothelial Bladder Cancer in the Upper-Urinary Tract
* Prostate or bladder radiotherapy
* Urinary tract infection
* Chronic urinary retention or indwelling catheters
* Other ongoing oncological diseases
* Active oncological treatments in the past 12 months
* Persistent disease (defined as residual disease detected within three months after TURB or at first cystoscopy)
* Specific dietary restrictions such as a vegetarian diet, celiac disease, or lactose intolerance
* Chronic Kidney Disease
* Chronic inflammatory diseases such as Crohn's disease or ulcerative colitis
* History of gastric resection
* Hepatic disorders such as cirrhosis or ALT/AST levels three times above the upper normal limit
* Thyroid disorders
* Warfarin therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-10-17 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence Free Survival | 24 months
  of recurrence-free survival (RFS) at 1 year, of a dietary regimen characterized by high consumption of the Cruciferae family vegetables versus no dietary regimen in patients with Intermediate, High, or Very High-grade Non-Muscle Invasive Bladder Cancer treated with BCG (defined as the standard of care - SOC).

SECONDARY OUTCOMES:
Recurrence in BCa | 24 months
  Recurrence, of a dietary regimen characterized by high consumption of the Cruciferae family vegetables versus no dietary regimen in patients with Intermediate, High, and Very High-grade Non-Muscle Invasive Bladder Cancer
ITC levels | 24 months
  To evaluate the impact of high Cruciferous vegetable consumption on urinary ITC levels.

CONTACTS AND LOCATIONS:
Overall Officials: Cosimo De Nunzio, Professor, Principal Investigator — Sant'Andrea Hospital of Rome
Locations (1):
- S.Andrea Hospital of Rome, Rome, Lazio, Italy

IPD SHARING:
Plan to Share IPD: Yes
Results will be published in an original article
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Two years

REFERENCES:
- See also: Burger M, Catto JWF, Dalbagni G, Grossman HB, Herr H, Karakiewicz P, Kassouf W, Kiemeney LA, La Vecchia C, Shariat S, Lotan Y. Epidemiology and risk factors of urothelial bladder cancer. Eur Urol [Internet]. 2013 [cited 2025 Jan 26];63(2):234-41. — https://pubmed.ncbi.nlm.nih.gov/22877502/
- See also: Egbers L, Grotenhuis AJ, Aben KK, Witjes JA, Kiemeney LA, Vermeulen SH. The prognostic value of family history among patients with urinary bladder cancer. Int J Cancer [Internet]. 2015 Mar 1 [cited 2025 Jan 26];136(5):1117-24 — https://pubmed.ncbi.nlm.nih.gov/24978702/
- See also: Jubber I, Ong S, Bukavina L, Black PC, Compérat E, Kamat AM, Kiemeney L, Lawrentschuk N, Lerner SP, Meeks JJ, Moch H, Necchi A, Panebianco V, Sridhar SS, Znaor A, Catto JWF, Cumberbatch MG. Epidemiology of Bladder Cancer in 2023: A Systematic Review of R — https://pubmed.ncbi.nlm.nih.gov/37198015/

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-09-13): https://cdn.clinicaltrials.gov/large-docs/37/NCT07391137/Prot_SAP_ICF_000.pdf